CLINICAL TRIAL: NCT04891874
Title: Adjuvant Stereotactic Body Radiation for Hepatocellular Carcinoma With Microvascular Invasion and Narrow Resection Margin
Brief Title: Adjuvant Radiotherapy for Resected Hepatocellular Carcinoma With MVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Changying Shi, Principal Investigator, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eastern HSH
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Stereotactic body radiotherapy; Micro vascular invasion; Narrow resection margin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Adjuvant SBRT after surgery group vs. surgery alone group.
Who Masked: Outcomes Assessor

ARMS (2):
- SBRT group (Experimental): Participants in SBRT group will receive SBRT as adjuvant radiotherapy for hepatocellular carcinoma with microvascular invasion and narrow resection margin.
  Interventions: Radiation: Stereotactic radiotherapy
- Surgery alone group (No Intervention): Participants in surgery alone group will not receive any adjuvant therapy after surgery for hepatocellular carcinoma.

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Radiation using stereotactic radiotherapy device.
  Arms: SBRT group

SUMMARY:
Positive micro vascular invasion in early stage hepatocellular carcinoma(HCC) leads to early recurrence after surgery. Adjuvant external radiotherapy will be applied in those patients to see if disease free survival and overall survival could be approved.

DETAILED DESCRIPTION:
Hepatocellular carcinoma(HCC) ranks the 6th most common cancer and is the 2nd leading cause of cancer-related death globally. Surgical resection remains the most efficient therapy in early stage. Though an anatomical resection of tumor lead to an up to 70% 5-year overall survival, the existence of micro vascular invasion(MVI) caused early recurrence. Stereotactic body radiation therapy (SBRT) has been proved to be efficient in treating vascular tumor thrombosis. The investigators tried to implement this technique in adjuvant setting for HCC after surgery with MVI. Participants with early stage HCC whose tumor locates closely to the main intrahepatic vascular will be regarded as potentially-not-enough-surgical-margin candidates. Surgical resection will be carried out as scheduled and an additional silver clip will be put into the margin. Postoperative pathological examination will detect micro vascular invasion or daughter nodule. MVI-positive candidates will be eligible for enrollment. Eligible participants will be randomized to two groups, SBRT group and surgery-alone(SA) group with 1-to-1 ratio. Participants in SBRT group will receive a 35Gy limited resection margin parenchyma SBRT after surgery, while participants in SA group just get surgery. Radiation related adverse events (AE) or reaction will be recorded and intervened necessarily. All participants will be followed up by investigators every three months. DFS, OS, and AEs are end points in this study.

ELIGIBILITY:
Inclusion Criteria:

1. solitary nodule;
2. tumor adjacent to the main trunk of hepatic vein, cava vena, or to the major branch of portal vein (including the lobar branch at least);
3. macro-vascular negative;
4. no previous treatment before surgery;
5. no previous hepatic surgery;
6. Child-Pugh score A for hepatic function.

Exclusion Criteria:

1. spontaneous rupture;
2. pathologically proved positive resection margin;
3. severe cirrhosis with hypersplenism or esophageal and gastric varices;
4. 4-weeks postoperative examination revealed α-fetal protein(AFP) still positive or new lesion in remnant liver;
5. postoperative complications required a secondary operation or more than 3 weeks'recovery from surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiamei Yang, MD, Principal Investigator — Secondary Military Medical Unversity, Shanghai
Locations (1):
- Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi C, Li Y, Geng L, Shen W, Sui C, Dai B, Lu J, Pan M, Yang J. Adjuvant stereotactic body radiotherapy after marginal resection for hepatocellular carcinoma with microvascular invasion: A randomised controlled trial. Eur J Cancer. 2022 May;166:176-184. doi: 10.1016/j.ejca.2022.02.012. Epub 2022 Mar 15. PMID 35303509

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBRT Group | Surgery Alone Group
Started | 38 (Participants in this period were recruited from August 1, 2015 to December 31, 2016.) | 38
Completed | 38 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBRT Group | Surgery Alone Group | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 69
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 33 | 32 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 38 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 38 | 38 | 76
Hepatitis Virus [Number; unit: Number of Participants With Hepatitis Vi] — The participants with hepatitis virus were recoreded in the baseline characteristics. Difference between the two groups in hepatitis will be examed.
  Number of Participants With Hepatitis Vi | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Participants Without Recurrence (Disease-free).
Description: Participants will be monitored for recurrence(disease) since enrollment. DFS was defined as time interval from randomization to the first recurrence. The unit of measure was month.
Time Frame: DFS rate at 5-years after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Group | Surgery Alone Group
Number analyzed (Participants) | 38 | 38
Participants | 16 | 28

2. Secondary Outcome: Overall Survival (OS) Rate.
Description: OS was defined as time interval from randomization to death.
Time Frame: OS rate at 5-years from randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Group | Surgery Alone Group
Number analyzed (Participants) | 38 | 38
Participants | 29 | 20

3. Other Pre Specified Outcome: Number of Participants Occured Adverse Events(AE)
Description: AE was defined as side effect related to the radiotherapy
Time Frame: AE will be evaluated up to 3 months after radiotherapy in SBRT group
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Group | Surgery Alone Group
Number analyzed (Participants) | 38 | 38
Participants | 12 | 0

ADVERSE EVENTS:
Time Frame: 3 months from radiotherapy.
Description: The adverse events were reported according to the CTCAE 5.0 version.
Groups:
- SBRT Group: Participants in SBRT group will receive SBRT as adjuvant radiotherapy for hepatocellular carcinoma with microvascular invasion and narrow resection margin. The AE like fatigue, vomitting, skin reaction and other items according to CTCAE5.0 will be recorded.
Arm/Group | SBRT Group | Surgery Alone Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 12/38 | 0/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT Group (N=38) | Surgery Alone Group (N=38)
Fatigue (General disorders) | 9 (9) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04891874/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04891874/SAP_001.pdf
  • Informed Consent Form (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04891874/ICF_002.pdf